CLINICAL TRIAL: NCT01615341
Title: Subclinical Viral Infection and Renal Allograft Injury
Brief Title: Study of Subclinical Viral Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Jodi Smith, Assistant Professor, Seattle Children's Hospital
Other Study IDs: R01DK088914-01A1 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Kidney Transplantation; Kidney Failure, Chronic
Keywords: Kidney transplantation; Subclinical Viral Infection; Renal Allograft Injury
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If participant agrees, blood, tissue, and study data will be banked at Seattle Children's Research Institute.
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic allograft injury is the leading cause of graft loss in renal transplantation. The shortage of available kidneys for transplantation has reached crisis levels with increasing numbers of waiting list mortalities. Strategies to prolong graft survival are urgently needed. The pediatric and young adult transplant population is one in which repeat transplantation is inevitable and therefore, this group is one who will especially benefit from intervention to prolong graft survival. The hypothesis of this proposal is that subclinical viral infection is a modifiable risk factor in the pathogenesis of chronic allograft injury. The young age of the proposed study population is an ideal one to evaluate this objective due to the high prevalence of seronegative recipients. The studies outlined will determine the temporal relationship betWeween subclinical viremia, renal allograft infection and allograft injury. This will be the first prospective study in renal transplant recipients to systematically monitor subclinical viral infection both in peripheral blood and in the renal allograft with concurrent quantitative measures of renal function, allograft fibrosis, and innate immune activation. The investigators have chosen these 3 outcomes because they evaluate a spectrum of renal allograft injury and represent different stages - from early to late - in the pathophysiology that leads to renal allograft dysfunction. In addition, the role of virus specific T cell immune responses in the control of subclinical viral infection and associated allograft injury will be determined. These data are critical as they will provide insights into the pathogenesis of injury and will guide development of interventions strategies. Importantly, the current treatment strategies for viral disease do not prevent subclinical viral infection. Thus, the results of this study may identify that prevention, prophylaxis and/or treatment of subclinical viral replication as a long term strategy to prevent chronic allograft injury and prolong graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent guardian must be able to understand and provide informed consent or assent
* Male or Female, Seattle Children's Hospital participants must be 1-<21 yrs and University of Washington Medical Center participants 18-25yrs.
* Diagnosed with End Stage Renal Disease (ESRD)

Exclusion Criteria:

* Inability or unwillingness of subject and/or parent guardian to provide informed consent
* Pregnancy

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and young adult renal transplant recipients (1<25yrs) of their first kidney transplant from Seattle Children's Hospital and University of Washington Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change in measured GFR from baseline | time of transplant, one time between months 3 and 6, and during months 12, and 24 after the transplant
  Single infusion of iohexol clearance to measure GFR

SECONDARY OUTCOMES:
Change in interstitial fibrosis and tubular atrophy of renal allograft from baseline | Renal biopsies will be performed at time of transplant, 3-6 m, 12m, and 24m post-transplant. Precise measures of renal function, allograft fibrosis, and innate immune activation will be performed at baseline, 6m, 12, 24m post-transplant.
Change in innate immune activation of renal allograft from baseline | 6, 12, and 24 months after the transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Smith, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States